CLINICAL TRIAL: NCT04308876
Title: Investigation of Effectiveness of Manual Therapy and Strengthening Exercises in Physiotherapy and Rehabilitation of Hemophilic Arthropathy of the Elbow
Brief Title: Effectiveness of Manual Therapy and Strengthening Exercises in Hemophilic Arthropathy of the Elbow Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Ayse Merve Tat, Lecturer, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Necmettin Erb. Physiotherapy-1
Record Dates: First submitted 2020-03-12; First posted 2020-03-16 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Hemophilia; Arthritis
Keywords: Hemophilia; Arthropathy; Elbow joint; Manual therapy; Exercise
MeSH Terms: conditions — Hemophilia A; Arthritis; Joint Diseases; Motor Activity | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual therapy and strengthening exercises (Experimental): Manual therapy and strengthening exercises were applied totally 15 sessions for 5 weeks 3 times a week in hospital by physiotherapist.
  Interventions: Other: Manual therapy; Other: Strengthening exercises
- Strengthening exercises (Active Comparator): Patients in this group performed the strengthening exercises given to the experimental group on their own at home with experimental group at the same time, frequency and dose.
  Interventions: Other: Strengthening exercises

INTERVENTIONS:
Other: Manual therapy — Manual therapy includes techniques applied to elbow joints and surrounding tissues
  Arms: Manual therapy and strengthening exercises
Other: Strengthening exercises — Strengthening exercises used in this study includes resistant exercises to increase muscle strength of upper extremity

SUMMARY:
Manual treatment involves techniques based on the principles of moving the joint faces and separating the joint gap, and soft tissues mobilization techniques. The use of manual therapy in hemophilia is gradually increasing although it previously described as a contraindication. The utility and use of strengthening exercises in hemophilia has been going on for a long time. In this study, the effect of manual therapy and strengthening exercises joint was investigated in hemophilic arthropathy of the elbow.

DETAILED DESCRIPTION:
The aim of this study was to investigate the effects of strengthening exercises and manual therapy on bleeding frequency, pain, range of motion, muscle strength, arm circumference, joint health, functionality and quality of life in the physiotherapy and rehabilitation of hemophilic arthropathy of the elbow. Seventeen adolescent and young adult hemophilic individuals aged 12-30 years with elbow arthropathy were included in the study. The individuals were divided into the two groups via simple randomisation as Manuel Therapy and Exercise Group (MTEG) and Home Exercise Group (HEG). The individuals in HEG were given strengthening exercises as a home program. Those in the MTEG were applied manual therapy by the physiotherapist and were given supervised strengthening exercises. All treatments were performed 3 times a week for 5 weeks totally 15 sessions. Frequency of bleeding was evaluated with number of bleeding in the last 5 weeks. Numerical Pain Scale was used for activity and resting pain. Range of motion and muscle strength were measured with universal goniometer and digital dynamometer, respectively. The Quick-DASH questionnaire and Oxford Elbow Score were used for the functionality of the upper extremity and quality of life, respectively. The joint health status was evaluated with Hemophilia Joint Health Score-Elbow Point and Hospital for Special Surgery-Elbow Scoring System. Evaluations were made by the same physiotherapist before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Having signs of hemophilic arthropathy in one or both elbow joints, Being between the ages of 12-30 (Adolescent and young adult), Receiving prophylactic factor replacement therapy.

Exclusion Criteria:

* Having undergone any surgical procedure for elbow arthropathy, Having an orthopedic problem, such as a fracture, ligament or tendon injury, related to the upper limb in the past year, Receiving physiotherapy and rehabilitation for the elbow joint in the last 6 months

Ages: 12 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2018-04-09 (Actual); Primary Completion 2019-03-10 (Actual); Study Completion 2020-02-06 (Actual)

PRIMARY OUTCOMES:
Hemophilia Joint Health Score | 5 week
  We used the elbow point of Joint Health Status. Elbow Point is scored 0-20. A high score indicates that arthropathy findings worsen
Frequency of bleeding | 5 week
  It was evaluated wit bleeding number in elbow joint over last 5 week
Numerical Pain Scale | 5 week
  It was used for evaluation of activity and resting pain.

SECONDARY OUTCOMES:
Range of motion | 5 week
  It was measured with universal goniometer.
Muscle strength | 5 week
  It was measured with digital dynamometer (Lafayette hand-held dynamometer)
Functionality of the upper extremity | 5 week
  Quick-Disability of Arm, Shoulder and Hand questionnaire was used.
Oxford Elbow Score | 5 week
  It was used for evaluation of Quality of life.
Physical status of the elbow | 5 week
  Hospital for Special Surgery-Elbow Scoring System was used.

CONTACTS AND LOCATIONS:
Overall Officials: Filiz Can, Professor, Study Chair — Hacettepe University, Faculty of Physical Therapy; Ilgen Sasmaz, Study Director — Cukurova University, Faculty of Medicine, Department of Pediatric Hematology
Locations (1):
- Cukurova University, Adana, Sarıcam, Turkey (Türkiye)